CLINICAL TRIAL: NCT00708721
Title: Phase I/II Study of Low-dose Oral Clofarabine for the Treatment of IPSS INT-1, INT-2 or HIGH Myelodysplastic Syndromes and Chronic Myelomonocytic Leukemia (Dysplastic Type) Patients Who Have Failed Hypomethylating Therapy
Brief Title: Low-dose Oral Clofarabine for the Treatment of IPSS INT-1, INT-2 or HIGH Myelodysplastic Syndromes and Chronic Myelomonocytic Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Data analysis revealed sufficient data for safety and efficacy
Sponsor: University of Utah (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI26135
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Cancer; Chronic Myelomonocytic Leukemia
Keywords: hypomethylating therapy; CML; myelodysplastic syndromes
MeSH Terms: conditions — Neoplasms; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental): All participants enrolled.
  Interventions: Drug: Clofarabine

INTERVENTIONS:
Drug: Clofarabine — Clofarabine is a rationally designed, second generation purine nucleoside analogue. Clofarabine was designed as a hybrid molecule to overcome the limitations and incorporate the best qualities of both fludarabine (F-ara-A) and cladribine (2-CdA, CdA) both of which are currently approved by various regulatory authorities for treatment of hematologic malignancies.
  Other Names: Clofarabine (2-chloro-9-[2-deoxy-2-fluoro-D-arabinofuranosyl]adenine; Cl-F-ara A; CAFdA

SUMMARY:
Study and Dose Rationale The safety profile of clofarabine appears acceptable within the target populations studied to date in the clinical studies summarized in Section 2.3. clofarabine has demonstrated anti-cancer activity through inhibition of DNA synthesis and repair, induction of apoptosis, and possibly through other mechanisms. The effect of clofarabine on DNA methylation has not been determined. Numerous responses have been observed after treatment with clofarabine in heavily pre-treated relapsed/refractory patients with ALL or AML.

Recently 2 small studies were conducted at the M.D. Anderson Cancer Center looking at the use of clofarabine in the treatment of MDS.31 The first study randomized patients in a Bayesian fashion to 15 vs. 30 mg/m2 given IV daily for 5 days every 4 to 8 weeks. In the 15 mg/m2 arm 3 of 7 patients had a complete remission according to the International Working Group (IWG)32 criteria for response. In the 30 mg/m2 arm, 2 of 6 patients had a complete remission while 1 patient had hematologic improvement according to IWG criteria. In the second study, patients were treated with oral clofarabine at a dose of 40 mg/m2 daily for 5 days every 4 to 8 weeks. Two of 7 patients had hematologic improvement according to IWG criteria. The main toxicities in both trials were prolonged myelosuppression and liver function abnormalities.

Preclinical animal models have shown increased clofarabine activity against multiple different tumors with repetitive daily dosing for prolonged periods of time.33 The use of an oral therapy is advantageous for the treatment of a chronic malignancy such as MDS. Furthermore, based on the pre-clinical data mentioned above daily repetitive dosing over a protracted period may provide increased efficacy. Since most MDS patients are elderly and may not tolerate aggressive therapy, a schedule of administration of low dose oral clofarabine over a protracted period may provide the advantage of increased efficacy without severe toxicity. The safety of a protracted daily dosage of oral clofarabine in humans has not been determined. The dosing scheme for this study will therefore include a dose escalating phase I component followed by a phase II component. The starting dose will be 5 mg (fixed dose) orally daily for 10 days. This dose will be escalated in cohorts of 3 patients as tolerated up to a maximal dose of 15 mg (fixed dose) orally for 10 consecutive days. Note that at the latter dose a patient will receive a total of 150 mg of clofarabine per cycle, which far lower than the MD Anderson study of oral clofarabine in MDS whereby patients received 200 mg/m2 per cycle.

OBJECTIVES:

Study Overview The purpose of this study is to determine the efficacy and toxicity of Clofarabine administered orally at a low daily dose for the treatment of myelodysplastic syndromes.

DETAILED DESCRIPTION:
Primary Objectives

1. Phase I: To determine the MTD within the planned dose range for this patient population and assess the toxicity of oral clofarabine
2. Phase II: To estimate the overall response rate (complete, partial and hematologic improvement by modified IWG criteria) in response to low dose daily oral clofarabine in patients with high risk myelodysplastic syndrome or chronic myelomonocytic leukemia (dysplastic type).

Secondary Objectives

1. To evaluate the toxicity of low dose daily oral clofarabine in this patient population.
2. To determine the time to progression to acute myeloid leukemia (AML) of MDS patients treated with low dose daily oral clofarabine.
3. To determine the duration of response, overall survival (OS) and progression free survival (PFS) of MDS patients treated with low dose daily oral clofarabine.
4. To determine the effect of low dose daily oral clofarabine on global methylation in patients with MDS.
5. To determine the effect of low dose daily oral clofarabine on miRNA and mRNA expression patterns in patients with MDS.

Treatment Patients will take Clofarabine by mouth once daily for 10 days followed by 18 days of no Clofarabine. This 28 day period of time is called one treatment cycle. After they complete three cycles of treatment they will have bone marrow and blood tests done to find out if their MDS or CMML is responding to the treatment. If these tests show the MDS or CMML is responding to treatment they will continue taking the same dose of Clofarabine for 3 more cycles. If the tests show that the MDS or CMML is not responding to treatment the dose of Clofarabine will be increased and they will continue on the same schedule (10 days on, 18 days off) for 3 more cycles.

After 6 cycles patients will again have bone marrow and blood tests done to find out if the MDS or CMML is responding to the treatment. If the tests show that the MDS or CMML is not responding to treatment the dose of Clofarabine will be increased again and they will continue on the same schedule (10 days on, 18 days off) for 6 more cycles.

5-3-11 Update: The phase I portion of the study has now been closed to accrual. The Phase II portion of the trial will enroll up to 20 patients. Patients will be evaluated on a weekly basis for toxicity. At the completion of cycle 3 and within 1 week of starting cycle 4, patients will receive a bone marrow aspirate and biopsy in addition to a complete blood count in order to evaluate for response according to IWG criteria. Patients who have evidence of a response to therapy or stable disease will be continued on the same dose and schedule of oral clofarabine. Bone marrow evaluation for response will be obtained at the completion of 6 and then 12 cycles. If the patient continues treatment after cycle 12 a bone marrow evaluation will be done at the discretion of the investigator. Treatment will continue at the same dose and schedule indefinitely until either disease progression, the development of unacceptable toxicity or the patient decides to go off study.

Follow-up For this protocol, all patients, including those who discontinue protocol therapy early, will be followed for response until progression and for survival for 5 years from the date of registration. All patients must also be followed through completion of all protocol therapy.

ELIGIBILITY:
Inclusion Criteria:

A bone marrow biopsy confirmed diagnosis of MDS or CMML (dysplastic subtype) according to WHO criteria within 2 weeks of registration.

1. Patients must have an International Prognostic Scoring System (IPSS), see Appendix D, score of INT-1 or higher at study entry.35 Patients with an IPSS score of INT-1 with the 5q- deletion should have failed Lenalidomide therapy and should have more than 5% blasts in the bone marrow or a platelet count < 50,000/mm3 or an absolute neutrophil count < 500/mm3 or be requiring therapy (e.g. being transfusion dependent). Patients with CMML must have a WBC < 12,000/mm3 documented within 4 weeks prior to study entry (two sets of counts that are 2 weeks apart will be taken).
2. Patients with MDS should have failed or relapsed after treatment with one regimen of hypomethylating agents (5-Azacytidine or Decitabine) but no more than 2 prior therapies including only 1 hypomethylating agent... Patients with CMML (dysplastic subtype) may be enrolled even if they have not received any prior therapy.
3. Untreated patients who are ineligible for or unwilling to undergo hypomethylating agent therapy can be enrolled
4. Age ≥ 18 years.
5. Patients must have and ECOG performance status of 0 - 2.
6. Provide signed written informed consent.
7. Have adequate renal and hepatic functions as indicated by the following laboratory values:

   * Serum creatinine 1.0 mg/dL; if serum creatinine 1.0 mg/dL, then the estimated glomerular filtration rate (GFR) must be 30 mL/min/1.73 m2 as calculated by the Modification of Diet in Renal Disease equation where Predicted GFR (ml/min/1.73 m2) = 186 x (Serum Creatinine)-1.154 x (age in years)-0.023 x (0.742 if patient is female) x (1.212 if patient is black)
   * Serum bilirubin ≤1.5 mg/dL × upper limit of normal (ULN)
   * Aspartate transaminase (AST)/alanine transaminase (ALT) 2.5 × ULN
   * Alkaline phosphatase 2.5 × ULN
8. Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent.
9. Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment.
10. Male and female patients must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment

Exclusion Criteria:

1. Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol.
2. Pre-treatment with more than 2 previous regimens.
3. Use of investigational agents within 30 days or any anticancer therapy within 30 days before study entry with the exception of hydroxyurea. The patient must have recovered from all acute toxicities from any previous therapy.
4. Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo treatment.
5. Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
6. Pregnant or lactating patients.
7. Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Shami, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: 5 mg/Day for 10 Days: 5 mg/day for 10 out of 28 days
- Cohort 2: 1 mg/Day for 10 Days: 1 mg/day for 10/28 days and for cycle 1 and then 1 mg/day for 7/28 days for cycle 2 onward
- Cohort 3: 1 mg/Day for 7 Days: 1 mg/day for 7/28 days
Period: Overall Study
Arm/Group | Cohort 1: 5 mg/Day for 10 Days | Cohort 2: 1 mg/Day for 10 Days | Cohort 3: 1 mg/Day for 7 Days | Not Evaluable
Started | 2 | 4 | 3 | 2
Completed | 2 | 4 | 3 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Groups
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 7
Age, Continuous [Mean (Full Range); unit: years] | 68.3 [59 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Dose-Limiting Toxicity
Description: Dose-limiting toxicity was defined as any nonhematologic toxicity grade 3 or greater except for alopecia or nausea (which may be of grade 4 severity), or any grade 4 hematologic toxicity lasting more than 28 days after the last day of therapy.
Time Frame: 28 days after the first admistration of oral clofarabine
Population: 9 out of 11 participants were evaluable for this outcome.
Measure: Number; unit: participants who experienced a DLT
Arm/Group | Cohort 1: 10 mg/Day for 10 Days | Cohort 2: 1 mg/Day for 10 Days | Cohort 3: 1 mg/Day for 7 Days | Not Evaluable
Number analyzed (Participants) | 2 | 4 | 3 | 2
participants who experienced a DLT | 2 | 4 | 0 | 0
Statistical Analysis 1: Comparison: Cohort 1: 10 mg/Day for 10 Days vs Cohort 2: 1 mg/Day for 10 Days; Test type: Other; Maximum Tolerated Dose = 1 — Based on cytopenias observed at day 10 (Phase 1 trial only), and the Phase II dose was determined to be 1 mg per day for 7 consecutive days given on a 28 day cycle

2. Primary Outcome: The Overall Response Rate in Response to Low Dose Daily Oral Clofarabine in Patients With High Risk Myelodysplastic Syndrome or Chronic Myelomonocytic Leukemia (Dysplastic Type).
Description: Response rate was measured as complete, partial and hematologic improvement by modified IWG criteria. For complete remission the following must be present for four weeks in a bone marrow aspirate and biopsy: <5% myeloblasts, normal maturation of all cell lines, persisted dysplasia. Peripheral blood counts need to be hemoglobin >11 g/dL, neutrophils >1000/mm3, platelets>100000/mm3, blasts 0%. Partial remission requires all criteria for complete remission except blasts decreased by >50% over pretreatment. Stable disease is defined as failure to achieve at least partial remission, but no evidence of progression for > 8 weeks. Failure is defined as death during tre3atment or disease progression characterized by worsening of cytopenias, increase in percentage of bone marrow blasts, or progression to a more advanced MDS FAB subtype than pretreatment.
Time Frame: 4 weeks
Population: Two patients were not eligible for analysis.
Measure: Number; unit: participants who experienced a response
Groups:
- All Evaluable Patients: All participants enrolled.
  Clofarabine: Clofarabine is a rationally designed, second generation purine nucleoside analogue. Clofarabine was designed as a hybrid molecule to overcome the limitations and incorporate the best qualities of both fludarabine (F-ara-A) and cladribine (2-CdA, CdA) both of which are currently approved by various regulatory authorities for treatment of hematologic malignancies.
Arm/Group | All Evaluable Patients
Number analyzed (Participants) | 9
participants who experienced a response | 3

3. Secondary Outcome: Time to Progression to Acute Myeloid Leukemia (AML)
Description: Longest documented duration of time until progression to AML.
Time Frame: approximately 4 years
Population: Cycles are 28 days long. Analysis assessed the longest number of cycles completed on study until progression to AML.
Measure: Number; unit: cycles
Groups:
- All Evaluable Patients: Only nine of the eleven patients were evaluable for this outcome measure.
Arm/Group | All Evaluable Patients
Number analyzed (Participants) | 9
cycles | 51

4. Secondary Outcome: Response of MDS Patients Treated With Low Dose Daily Oral Clofarabine.
Description: Stable disease is defined as failure to achieve at least PR, but no evidence of progression for > 8 weeks.
Time Frame: approximately 4 years
Population: Of 11 patients, 9 were evaluable for response. Two patients had stable disease responses.
Measure: Count of Participants; unit: Participants
Groups:
- All Evaluable Patients: All evaluable patients. Eleven patients were enrolled, but only nine were evaluable.
Arm/Group | All Evaluable Patients
Number analyzed (Participants) | 9
Participants | 2

5. Secondary Outcome: The Effect of Low Dose Daily Oral Clofarabine on Global Methylation in Patients With MDS.
Description: Potential genomic changes following low dose daily oral clofarabine administration will be assessed.
Time Frame: through end of treatment
Population: Data were not collected and the outcome measure was not analyzed
Arm/Group | All Patients
Number analyzed (Participants) | 0
Value | 0

6. Secondary Outcome: The Effect of Low Dose Daily Oral Clofarabine on miRNA and mRNA Expression Patterns in Patients With MDS
Description: Assessment of potential change in miRNA and mRNA genetic expression patterns in patients following administration of low dose daily clofarabine.
Time Frame: through end of treatment
Population: Data were not collected and the outcome measure was not analyzed
Arm/Group | All Patients
Number analyzed (Participants) | 0
Value | 0

7. Secondary Outcome: Number of Participants With Adverse Events
Description: NCI CTCAE version 3.0 will be used to assess adverse events. The number of participants experiencing adverse events and the number of adverse events per patient will be documented through the course of study.
Time Frame: To 30 days after end of treatment or until full resolution.
Population: All participants experienced at least 1 adverse event (100% of the patient population; 11/11 participants)
Measure: Number; unit: participants experiencing adverse events
Arm/Group | All Patients
Number analyzed (Participants) | 11
participants experiencing adverse events | 11

ADVERSE EVENTS:
Time Frame: Adverse events were collected after the administration of the study drug and followed until resolution.
Groups:
- All Groups: All patients who received study treatment.
Arm/Group | All Groups
Serious Adverse Events (participants affected / at risk) | 8/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Groups (N=11)
Subdural hematoma (Vascular disorders) | 1
pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
femur fracture (Musculoskeletal and connective tissue disorders) | 1
thrombocytopenia (Blood and lymphatic system disorders) | 2
cellulitis right forearm (Infections and infestations) | 1
urinary tract infection (Infections and infestations) | 1
cytopenia (Blood and lymphatic system disorders) | 1
febrile neutropenia (Blood and lymphatic system disorders) | 1
joint swelling (Musculoskeletal and connective tissue disorders) | 1
e. coli positive (Infections and infestations) | 1
Ovarian abscess (Reproductive system and breast disorders) | 1
mental status change (Nervous system disorders) | 1
congestive heart failure (Cardiac disorders) | 2
stroke (Nervous system disorders) | 1
gram positive cocci (Infections and infestations) | 1
renal failure (Renal and urinary disorders) | 1
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
cholecystitis (Gastrointestinal disorders) | 1
pulmonary hypertension (Cardiac disorders) | 1
decreased ejection fraction (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Groups (N=11)
allergic rhinits (Respiratory, thoracic and mediastinal disorders) | 1
anemia (Blood and lymphatic system disorders) | 7
leukopenia (Blood and lymphatic system disorders) | 4
lymphopenia (Blood and lymphatic system disorders) | 5
neutropenia (Blood and lymphatic system disorders) | 6
splenomegaly (Blood and lymphatic system disorders) | 1
thrombocytopenia (Blood and lymphatic system disorders) | 9
Afibrilation with RVR (Cardiac disorders) | 1
Atrial Flutter with AV Block (Cardiac disorders) | 1
Ventricular Tachycardia (Cardiac disorders) | 1
Cardiomegaly (Cardiac disorders) | 2
Hypertension (Cardiac disorders) | 1
Inferior Cardiac Infarct (Cardiac disorders) | 1
pericarditis (Cardiac disorders) | 1
elevated PTT (Cardiac disorders) | 1
diaphoretic (General disorders) | 1
fatigue (General disorders) | 7
fever (General disorders) | 3
insomnia (Psychiatric disorders) | 2
brusing (Injury, poisoning and procedural complications) | 3
cracked lips (Skin and subcutaneous tissue disorders) | 1
dry skin (Skin and subcutaneous tissue disorders) | 2
hernia (Injury, poisoning and procedural complications) | 1
itching (Skin and subcutaneous tissue disorders) | 1
lesions (Skin and subcutaneous tissue disorders) | 4
rash: erythemia (Skin and subcutaneous tissue disorders) | 3
ulceration (Skin and subcutaneous tissue disorders) | 2
hot flashes (Vascular disorders) | 1
vomiting (Gastrointestinal disorders) | 2
abdominal distention (Gastrointestinal disorders) | 1
abdominal pain (Gastrointestinal disorders) | 5
anorexia (Metabolism and nutrition disorders) | 4
blood blisters in mouth (Gastrointestinal disorders) | 1
constipation (Gastrointestinal disorders) | 2
diarrhea (Gastrointestinal disorders) | 3
flatulence (Gastrointestinal disorders) | 1
heart burn (Gastrointestinal disorders) | 1
mouth sores (Gastrointestinal disorders) | 1
nausea (Gastrointestinal disorders) | 4
oral thrush (Gastrointestinal disorders) | 2
hematomas (Blood and lymphatic system disorders) | 1
petechia (Blood and lymphatic system disorders) | 4
c. differential positive (Infections and infestations) | 1
cellulitis (Infections and infestations) | 1
eye infection (Infections and infestations) | 1
head cold (Infections and infestations) | 1
infections with unknown ANC (Infections and infestations) | 1
neutropenic fever (Blood and lymphatic system disorders) | 1
prostatitis (Infections and infestations) | 1
sepsis (Infections and infestations) | 1
sore throat (Infections and infestations) | 1
upper respiratory infection (Infections and infestations) | 2
yeast infection (Infections and infestations) | 1
edema (bilateral lower extremity) (General disorders) | 3
pedal edema (General disorders) | 1
elevated alkaline phosphatase (Investigations) | 3
elevated ALT (Investigations) | 2
elevated amylase (Investigations) | 1
elevated AST (Investigations) | 4
elevated uric acid (Metabolism and nutrition disorders) | 1
Hyperbilirubinemia (Investigations) | 3
hypercalcemia (Metabolism and nutrition disorders) | 1
hyperglycemia (Metabolism and nutrition disorders) | 7
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
hypocalcemia (Metabolism and nutrition disorders) | 2
hypoglycemia (Metabolism and nutrition disorders) | 3
hyponatremia (Metabolism and nutrition disorders) | 2
increased creatinine (Investigations) | 3
hypokelmia (Metabolism and nutrition disorders) | 2
bilateral leg weakness (Musculoskeletal and connective tissue disorders) | 1
fracture (Musculoskeletal and connective tissue disorders) | 2
hand laceration (Musculoskeletal and connective tissue disorders) | 1
muscle cramps (Musculoskeletal and connective tissue disorders) | 1
muscle weakness (Musculoskeletal and connective tissue disorders) | 1
confusion (Nervous system disorders) | 2
dizziness (Nervous system disorders) | 3
drowsiness (Nervous system disorders) | 1
hallucination (Nervous system disorders) | 1
neuropathy: cranial (Nervous system disorders) | 1
neuropathy: motor (Nervous system disorders) | 1
anxiety (Nervous system disorders) | 2
syncope (Nervous system disorders) | 1
left eye redness (Eye disorders) | 1
eye scratch (Eye disorders) | 1
back pain (Musculoskeletal and connective tissue disorders) | 4
chest pain (General disorders) | 3
dysuria (Renal and urinary disorders) | 1
headache (Nervous system disorders) | 3
joint pain (Musculoskeletal and connective tissue disorders) | 1
oral pain (Gastrointestinal disorders) | 1
right knee pain (Musculoskeletal and connective tissue disorders) | 1
throat pain (Gastrointestinal disorders) | 1
pain at port site (General disorders) | 1
rib pain (Metabolism and nutrition disorders) | 1
atelectasis (Respiratory, thoracic and mediastinal disorders) | 2
bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
chest congestion (Respiratory, thoracic and mediastinal disorders) | 1
cough (Respiratory, thoracic and mediastinal disorders) | 5
crackles in lungs (Respiratory, thoracic and mediastinal disorders) | 1
Dyspenia (Respiratory, thoracic and mediastinal disorders) | 3
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
pneumonia (Respiratory, thoracic and mediastinal disorders) | 3
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
wheezing (Respiratory, thoracic and mediastinal disorders) | 1
lower extremity phlebitis (Vascular disorders) | 1
superficial thrombosis (Vascular disorders) | 1
pericardial thickening (Cardiac disorders) | 1
urinary tract infection (Infections and infestations) | 2
arthritis (Musculoskeletal and connective tissue disorders) | 1
bone pain (Musculoskeletal and connective tissue disorders) | 1
bleeding in mouth (Gastrointestinal disorders) | 1
night sweats (Skin and subcutaneous tissue disorders) | 1
erythematous (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No